CLINICAL TRIAL: NCT00709215
Title: A Phase I/II Study of Cordycepin Plus Pentostatin in Patients With Refractory TdT-Positive Leukemia
Brief Title: Study of Cordycepin Plus Pentostatin in Patients With Refractory TdT-Positive Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: OncoVista, Inc. (Industry)
Collaborators: AAIPharma (Industry)
Responsible Party: Michael Moloney, Director - Program Management, OncoVista, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OV06-001
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Refractory TdT-Positive Leukemia
Keywords: refractory TdT-positive leukemia; ALL; AML; blastic CML
MeSH Terms: interventions — cordycepin; Pentostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cordycepin plus Pentostatin — Cordycepin Plus Pentostatin on days 1, 2 and 3 of a 21 day cycle. Number of cycles until progression or unacceptable toxicity

SUMMARY:
This is a two-part, open-label, Phase I/II study in subjects with relapsed or refractory TdT-positive leukemia for which no standard therapies are expected to result in durable remission.

DETAILED DESCRIPTION:
In the first phase the Study Objectives are to:

* Define the maximally tolerated dose (MTD) and recommended dose (RD) for administration of cordycepin as a 1-hour IV infusion, administered 1 hour following administration of an IV bolus of pentostatin, in subjects with refractory TdT-positive leukemia;
* Determine plasma ADA levels prior to pentostatin infusion and at 60 and 120 minutes after administration of pentostatin;
* Determine the single and multiple dose pharmacokinetics (PK) of cordycepin given 1 hour after a fixed dose of pentostatin;
* Assess cordycepin pharmacodynamics by measurement of blast cell apoptosis from peripheral blood smears;
* Measure and quantitate any clinical responses in refractory TdT-positive leukemia patients following cordycepin/pentostatin administration.

In the second phase, the Study Objectives are to assess the safety, PK, and clinical outcomes of cordycepin in combination with pentostatin, at the RD, in a 20 subject cohort

ELIGIBILITY:
Inclusion Criteria:

* TdT-positive leukemia (ALL, AML, or blastic CML) that has failed at least one standard treatment regimen and for which no standard therapies are expected to result in durable remission. Leukemia is minimally defined as at least 20% blast cells present in marrow or peripheral blood. TdT must be expressed in at least 20% of blast cells present and documented either immunologically or biochemically;
* Age ≥18 years;
* Must understand and voluntarily sign informed consent;
* Adequate non-hematologic organ system function, defined by:

  * Creatinine ≤1.5 times the upper limit of normal (ULN) and/or creatinine clearance ≥60 mL/min
  * AST and/or ALT ≤2.5 times upper limit of normal (ULN)
  * Total bilirubin within institutional normal range
  * Normal EKG and LVEF >40%, measured by EKG and MUGA scan, radionuclide ventriculogram, or echocardiogram
* Life expectancy >3 months;
* Performance status (PS) >70% Karnofsky or ECOG ≤2;
* Women of childbearing potential must have a negative serum pregnancy test within 7 days of starting study drug. A woman of child-bearing potential is a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e., who has had menses at any time in the preceding 24 consecutive months);
* Male or female of child-bearing potential must agree to use adequate contraceptive methods

Exclusion Criteria:

* Failure to meet inclusion criteria;
* Uncontrolled active infection;
* Extramedullary (CNS) disease;
* Serious concomitant medical illness, such as active infection, uncontrolled congestive heart failure, or uncontrolled diabetes or other metabolic disorder, or psychiatric illness;
* Pregnancy or lactation; females of child bearing potential must use adequate contraceptive methods;
* Less than 3 weeks since prior chemotherapy, radiation therapy, or immunotherapy. However, hydroxyurea is permitted up to 24 hours before the study is initiated;
* Less than 2 months following bone marrow or peripheral blood stem cell transplantation or treatment with donor lymphocyte infusion (DLI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Establishment of the recommended dose (RD) of cordycepin, given one hour following a fixed dose of the ADA inhibitor pentostatin, in subjects with refractory TdT-positive leukemia | one year

SECONDARY OUTCOMES:
Determination of the single and multiple dose pharmacokinetics of cordycepin. Measurement and quantification any any clinical responses following administration of cordycepin/pentostatin at the recomme | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Swaminathan Padmanabhan, MD, Principal Investigator — Cancer Therapy Research Center at UTHSCSA; Daneil J DeAngelo, MD, PhD., Principal Investigator — Dana Farber Cancr Institute
Locations (3):
- United States (3):
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Therapy Reasearch Center at UTHSCA, San Antonio, Texas

REFERENCES:
- [Derived] Verma AK. Cordycepin: a bioactive metabolite of Cordyceps militaris and polyadenylation inhibitor with therapeutic potential against COVID-19. J Biomol Struct Dyn. 2022 May;40(8):3745-3752. doi: 10.1080/07391102.2020.1850352. Epub 2020 Nov 23. PMID 33225826